CLINICAL TRIAL: NCT06458387
Title: Comparison of Clinical Outcomes According to High-protein Provision Through Parenteral Nutrition in Critically Ill Patients Immediately After Abdominal Surgery: a Prospective, Single-blinded, Randomized Controlled Trial
Brief Title: Comparison of Clinical Outcomes According to High-protein Provision in Critically Ill Patients After Abdominal Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Eun Young Kim, Professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SeoulSt_HP_01
Record Dates: First submitted 2024-06-05; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Protein Malnutrition
MeSH Terms: conditions — Kwashiorkor

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active protein supplementation (Experimental): The participants in active nutritional supplementation arm received nutritional support targeting specific protein (over 1.5 g/kg/day), with consultation from the nutritional support team and the initiation of nutritional supplementation on the same day as intensive care unit admission.
  Interventions: Dietary Supplement: Active protein supplementation
- Conventional protein supplementation (Experimental): The participants in conventional protein supplementation arm underwent conventional nutrition management without specific protein targets, but less than 1.5 g/kg/day.
  Interventions: Dietary Supplement: Conventional protein supplementation

INTERVENTIONS:
Dietary Supplement: Active protein supplementation — The participants in active nutritional supplementation arm received consultation from the nutritional support team (NST) upon ICU admission, and nutritional supplementation was initiated on the same day. NST is a multidisciplinary support team comprised of physicians, nurses, dietitians, and pharmacists, which assesses the nutritional status of patients, and provides recommendations for nutritional therapy. Targets in the participants in active protein supplementation arm were protein supplementation at over 1.5 g/kg/day during first 3 days after ICU admission. Actual body weight was used as the body weight for patients with a percent of ideal body weight (PIBW) of less than 120%, while adjusted body weight was used for patients with a PIBW greater than or equal to 120%.
  Arms: Active protein supplementation
Dietary Supplement: Conventional protein supplementation — The participants in conventional protein supplementation arm received conservative nutritional management without specific protein targets.
  Arms: Conventional protein supplementation

SUMMARY:
Protein malnutrition in critically ill patients is a global concern due to its association with prolonged hospital stays, and higher morbidity rates. Patients who undergo abdominal surgery are particularly vulnerable due to alterations in gastrointestinal function and prolonged fasting. Despite the significance of proper nutrition, the optimal target of protein supplementation remains controversial.

The investigators aimed to evaluate the effects of high protein provision, targeting a protein intake of at least 1.5 g/kg/day for the first 3 days after abdominal surgery, on 6-month mortality.

DETAILED DESCRIPTION:
During the acute phase of critical illness, patients experience metabolic and physiological changes that affects their nutrition status. One prominent feature is the activation of stress hormones and inflammatory mediators, which contribute to a negative nitrogen balance, increased gluconeogenesis, and accelerated muscle proteolysis. Among these patients, those who undergo abdominal surgery are particularly vulnerable to malnutrition as they experience alterations in the structural barrier of the gastrointestinal tract, impaired nutrient absorption, and prolonged fasting due to concerns such as the integrity of an anastomosis. Thus, appropriate protein provision should be prioritized for critically ill patients following abdominal surgery, and it should include adequate nutritional support to preserve lean body mass and organ function. Despite the importance of nutritional supply, the recommendations for protein vary according to different guidelines, and this is the same for surgical patients. Recent randomized controlled trials reported conflicting results with current guidelines, with some suggesting that higher protein dose administrations did not significantly impact clinical outcomes and may even worsen the outcomes for certain patient groups. Thus, the optimal protein provision target during the acute phase of critical illness, particularly for surgical patients, remains controversial.

The investigators aimed to assess the effects of strict high protein provision between the high protein group (protein target supplemented with 1.5 g/kg/day) and the control group (protein target supplemented with less than 1.5 g/kg/day) using intravenous nutrient solution for the first 3 days after abdominal surgery. Additionally, the investigators investigated the appropriate target for protein provision in critically ill patients who undergo abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted after abdominal surgery to our institution's surgical ICU
* They were enrolled regardless of the surgical method, either open, laparoscopy, or robotic.

Exclusion Criteria:

* aged under 18 years
* underwent surgery under local or regional anesthesia
* pregnant
* readmitted to the ICU due to any cause
* diagnosed with renal failure and receiving renal replacement therapy
* patients diagnosed with multiorgan failure, represented by a high Sequential Organ Failure Assessment (SOFA) score (≥9) upon ICU admission
* failed to provide informed consent, or with 'do-not-resuscitate' status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
6-month mortality rate | Participants were followed up to 180 days immediately after the surgery
  Proportion of patients who died within 6 months after surgery among participants

SECONDARY OUTCOMES:
30-day mortality rate | Participants were followed up to 30 days immediately after the surgery
  Proportion of patients who died within 30 days after surgery among participants
90-day mortality rate | Participants were followed up to 90 days immediately after the surgery
  Proportion of patients who died within 90 days after surgery among participants
Incidence of postoperative complications | Participants were followed during hospitalization (up to 14 days)
  Proportion of patients who developed any complications during postoperative hospitalization among participants

CONTACTS AND LOCATIONS:
Overall Officials: Hye sung Kim, Study Director — The Catholic University of Korea
Locations (1):
- Division of Trauma and Surgical Critical Care, Department of Surgery, Seoul St. Mary's Hospital, Seoul, Seocho-gu, Banpo-dong Banpodaero 222, South Korea